CLINICAL TRIAL: NCT00536224
Title: Brief Intervention to Promote Cardiovascular Risk Reduction in Patients Admitted to Chest Pain Observation Units
Brief Title: Chest Pain Observation Unit Risk Reduction Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: David A Katz (Other)
Collaborators: American Heart Association (Other)
Responsible Party: Sponsor-Investigator, David A Katz, Associate Professor of Medicine, University of Iowa
Organization: University of Iowa (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 200702770
Record Dates: First submitted 2007-09-25; First posted 2007-09-27 (Estimated); Last update posted 2018-04-26 (Actual); Status verified 2018-04

CONDITIONS: Chest Pain
Keywords: Health promotion; Emergency Medical Services; Randomized controlled trial; Chest pain observation unit; Cardiovascular risk factors
MeSH Terms: conditions — Chest Pain

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 2 (Active Comparator): Minimal counseling
  Interventions: Behavioral: Minimal counseling
- 1 (Experimental): Full counseling
  Interventions: Behavioral: Full counseling

INTERVENTIONS:
Behavioral: Full counseling — The health educator generated a computerized report for the patient that outlined his/her Framingham risk score, the goal for each cardiovascular risk factor based on national guidelines, and recommended actions for achieving each goal. Based on the Ask-Advise-Assess-Assist-Arrange follow-up (5A's) framework for behavior change, counseling for specific risk-related behaviors (diet, physical activity, and smoking) was provided by a cardiovascular rehabilitation health educator in the emergency department and during telephone follow-up (2 sessions over 6 weeks). Patients also received a general informational handout on self-management of cardiovascular risk factors (AHA Brochure "Controlling your risk factors"). A full report was also be sent to the patient's primary care physician (if any) at the conclusion of counseling.
  Arms: 1
Behavioral: Minimal counseling — Patients assigned to the minimal counseling intervention received brief counseling (<5 minutes) on the benefits of changing lifestyle and a handout with general information on self-management of cardiovascular risk factors.
  Patients assigned to minimal intervention also received an AHA brochure ("Controlling your risk factors") with general information on management of cardiovascular risk factors. At the end of 6-month follow-up, patients received a computerized report that outlined their Framingham risk score, the goal for each cardiovascular risk factor based on national guidelines, and recommended actions for achieving each goal.
  Arms: 2

SUMMARY:
The purpose of this study is to determine whether a brief counseling intervention initiated in the chest pain observation unit has a significant impact upon the health attitudes (readiness to change) and cardiovascular risk-related behaviors (diet, exercise, and smoking) of emergency department patients.

DETAILED DESCRIPTION:
Increasingly, emergency department patients for whom a non-ischemic etiology of acute coronary syndrome (ACS) symptoms cannot be identified undergo further evaluation to rule out myocardial ischemia and appraisal of cardiovascular risk factors (CRFs) in chest pain observation units (CPOUs). CPOU admission may represent a "teachable moment," but there has been little research on the effectiveness of brief, practical interventions for cardiovascular risk reduction in this population, despite the fact that the vast majority of these patients have at least one modifiable CRF and many do not receive regular primary care follow-up. The purpose of this study is to determine whether a brief counseling intervention initiated in the CPOU has a significant impact upon health attitudes (readiness to change) and cardiovascular risk-related behaviors (diet, exercise, and smoking). Based on the Health Belief Model (HBM), the intervention is designed to provide patients with tailored information on their cardiovascular risk, to negotiate goals for change, and to build problem-solving skills. All participants who are admitted to the CPOU for evaluation of ACS symptoms will be randomized to brief intervention (face-to-face counseling in the CPOU, coupled with telephone counseling at 4 weeks) or to minimal intervention (booklet with general information on CRFs) after a negative initial troponin measurement. We will conduct a baseline survey and follow-up telephone interviews at 2- and 6-month to assess stage of change and CRF-related behaviors. Linear mixed models and logistic regression (with generalized estimating equations) will be used to compare continuous and dichotomous behavioral outcomes across treatment arms, respectively. The proposed trial will evaluate the feasibility and effectiveness of delivering brief interventions for cardiovascular risk reduction in the CPOU setting, will provide insight into mechanisms of behavior change in these patients, and will guide the development of future case management interventions.

ELIGIBILITY:
Inclusion Criteria:

* At least one modifiable cardiovascular risk factor (smoking, hyperlipidemia, hypertension, diabetes mellitus, obesity)

Exclusion Criteria:

* Patients who "rule-in" for myocardial ischemia at initial testing
* Terminally ill (expected to survive less than 3 months)
* Unavailable for 6-month follow-up
* Cannot be contacted by telephone
* Institutionalized persons (prisoners, nursing home residents)
* Unable to provide informed consent (impaired mental status, unable to speak English)

Ages: 30 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Actual)
Dates: Start 2007-09; Primary Completion 2009-07 (Actual); Study Completion 2017-01 (Actual)

PRIMARY OUTCOMES:
Stage of change for cardiovascular risk-related behaviors (diet, exercise, and smoking) | 2- and 6-months
Self-reported cardiovascular health behaviors (diet, physical activity, and smoking cessation) | 2- and 6-months

CONTACTS AND LOCATIONS:
Overall Officials: David A Katz, MD, MSc, Principal Investigator — University of Iowa
Locations (1):
- University of Iowa Hospital, Iowa City, Iowa, United States

REFERENCES:
- [Background] Katz DA, Graber M, Birrer E, Lounsbury P, Baldwin A, Hillis SL, Christensen AJ. Health beliefs toward cardiovascular risk reduction in patients admitted to chest pain observation units. Acad Emerg Med. 2009 May;16(5):379-87. doi: 10.1111/j.1553-2712.2009.00383.x. Epub 2009 Mar 16. PMID 19302365
- [Result] Katz DA, Graber M, Lounsbury P, Vander Weg MW, Phillips EK, Clair C, Horwitz PA, Cai X, Christensen AJ. Multiple Risk Factor Counseling to Promote Heart-healthy Lifestyles in the Chest Pain Observation Unit: Pilot Randomized Controlled Trial. Acad Emerg Med. 2017 Aug;24(8):968-982. doi: 10.1111/acem.13231. Epub 2017 Jul 29. PMID 28748625